CLINICAL TRIAL: NCT05659446
Title: Endoscopic Management Of Low Output Recurrent Colonic Fistula Or Leak After Anterior Resection For Rectal Cancer: A Randomized Controlled Trial.
Brief Title: Endoscopic Management Of Low Output Recurrent Colonic Fistula Or Leak After Anterior Resection For Rectal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Said Mohamed Said Abdou Negm, lecturer of general surgery, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Amr Fouad
Record Dates: First submitted 2022-12-13; First posted 2022-12-21 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Colonic Fistula
Keywords: colonic fistula , endoscopy, leak, cancer rectum ,endoclip

STUDY DESIGN:
Intervention Model Description: This prospective randomized controlled clinical trial included all patients who developed the manifestations of low output recurrent colonic fistula or leak after colonic anterior resection for rectal cancer at Zagazig University hospital between (December 2020 to August 2022). the calculated sample size equal 78 patients divided into two equal groups.endoscopicgroup included 39 patients and surgical group included 39 patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- endoscopic group (Active Comparator): Patients involved in endoscopic group were firstly subjected for Interventional Radiology to drain any intra-peritoneal collection present in preoperative radiology then were subjected either to Clips application (OTSC, OVASCO Endoscopy AG. Tubingen, Germany) or Endo-suturing (Overstitch, Apollo Endo-Surgery , TX, United states) to close the low output fistula or leak after anterior resection for rectal cancer. The endoscopy was done under sedation, not general anesthesia after colonic preparation (chemical & mechanical preparation) firstly, to detect size of fistula . Clips were used in cases with fistula's size less than 10 mm, while Endo-suturing devices were used in cases with fistula's size more than 10mm till 15mm.
  Interventions: Procedure: endoscopy management of low output colonic fistula or leak after anterior resection for rectal cancer
- surgical group (No Intervention): Patients involved in surgical group were subjected to either redo of resection anastomosis manually or by circular stapler or primary repair of the defect with ileostomy. This was done under general anesthesia after colonic preparation.

INTERVENTIONS:
Procedure: endoscopy management of low output colonic fistula or leak after anterior resection for rectal cancer — Patients involved in endoscopic group were firstly subjected for Interventional Radiology to drain any intra-peritoneal collection present in preoperative radiology then were subjected either to Clips application (OTSC, OVASCO Endoscopy AG. Tubingen, Germany) or Endo-suturing (Overstitch, Apollo Endo-Surgery , TX, United states) to close the low output fistula or leak after anterior resection for rectal cancer. The endoscopy was done under sedation, not general anesthesia after colonic preparation (chemical & mechanical preparation) firstly, to detect size of fistula . Clips were used in cases with fistula's size less than 10 mm, while Endo-suturing devices were used in cases with fistula's size more than 10mm till 15mm.
  Arms: endoscopic group

SUMMARY:
This prospective randomized controlled clinical trial included all patients who developed the manifestations of low output recurrent colonic fistula or leak after colonic anterior resection for rectal cancer at Zagazig University hospital between (December 2020 to August 2022). The study was prospectively approved by Zagazig University Faculty of Medicine Institutional Review Board (Approval Number: 10027/26-10-2022) .The investigators performed the study under the code of ethics of the World Medical Association (Declaration of Helsinki) for studies involving human subjects. They got written informed consent from all participants after explaining to them all the study procedures with its benefits and hazards. Patients with recurrent low output colo-cutaneous fistula (less than 500cc/24h) or leak after anterior resection due to rectal cancer , patients who subjected to conservative measures but failed , patient with good general condition (ASA I&II), patients with size of fistula less than 15mm and patients with good nutritional status were included and eligible for randomization. The investigators excluded patients who were with bad general condition (ASAIII&IV&V), patients with high output fistula , patients with recto-vaginal or recto-vesical fistula, patients with size of fistula more than 15mm and patients were treated with conservative measures.

Included eligible patients were simply randomized at a 1:1 ratio to "Endoscopic (SG)" or "Surgical Group (EG)" via the drawing of sealed envelopes containing computer-generated random numbers prepared by a third party before the start of the intervention.

DETAILED DESCRIPTION:
This prospective randomized controlled clinical trial included all patients who developed the manifestations of low output recurrent colonic fistula or leak after colonic anterior resection for rectal cancer at Zagazig University hospital between (December 2020 to August 2022). The study was prospectively approved by Zagazig University Faculty of Medicine Institutional Review Board (Approval Number: 10027/26-10-2022).The investigators performed the study under the code of ethics of the World Medical Association (Declaration of Helsinki) for studies involving human subjects. They got written informed consent from all participants after explaining to them all the study procedures with its benefits and hazards. Patients with recurrent low output colo-cutaneous fistula (less than 500cc/24h) or leak after anterior resection due to rectal cancer , patients who subjected to conservative measures but failed , patient with good general condition (ASA I&II), patients with size of fistula less than 15mm and patients with good nutritional status were included and eligible for randomization. The investigators excluded patients who were with bad general condition (ASAIII&IV&V), patients with high output fistula , patients with recto-vaginal or recto-vesical fistula, patients with size of fistula more than 15mm and patients were treated with conservative measures.

Included eligible patients were simply randomized at a 1:1 ratio to "Endoscopic (SG)" or "Surgical Group (EG)" via the drawing of sealed envelopes containing computer-generated random numbers prepared by a third party before the start of the intervention.

The sample size was calculated by using an open Epi program depending on the following data; confidence interval 95%, power of the test 80%, ratio of unexposed/ exposed 1, the success rate of endoscopic management of low output colonic fistula after anterior resection of rectal cancer versus surgical management was 60.2% versus 90% respectively . Odd ratio 0.17, and risk ratio 0.67, so the calculated sample size equal 78 patients divided into two equal groups.

Primary and secondary outcomes were success rate in managing the fistula , postoperative hospital stay, and complications and mortality in each group after the intervention during the 3-months follow-up period, respectively.

Diagnosis After full history taking and complete physical examination, low output colonic fistula or leak after anterior resection for rectal cancer was clinically suspected and then confirmed by laboratory investigations (complete blood picture, liver and kidney functions, coagulation profile), radiological imaging (abdominal US to exclude any abdominal collection, CT abdomen with oral and I. V contrast, MRI in some situations and virtual colonoscopy to exclude any distal obstruction , distal narrowing or recurrence of the cancer ).

Intervention:

Patients involved in endoscopic group were firstly subjected for Interventional Radiology to drain any intra-peritoneal collection present in preoperative radiology then were subjected either to Clips application (OTSC, OVASCO Endoscopy AG. Tubingen, Germany) or Endo-suturing (Overstitch, Apollo Endo-Surgery , TX, United states) to close the low output fistula or leak after anterior resection for rectal cancer. The endoscopy was done under sedation, not general anesthesia after colonic preparation (chemical & mechanical preparation) firstly, to detect size of fistula . Clips were used in cases with fistula's size less than 10 mm, while Endo-suturing devices were used in cases with fistula's size more than 10mm till 15mm.

Patients involved in surgical group were subjected to either redo of resection anastomosis manually or by circular stapler or primary repair of the defect with ileostomy. This was done under general anesthesia after colonic preparation.

Follow up after endoscopy and discharge from the hospital:

All patients were subjected for clinical examination & laboratory investigation during the hospital stay. Any suspected colonic leak or fistula post intervention mandated CT scan with oral and I.V contrast and lower GI endoscopy. Patients were followed-up for at least 3 months post repair.

Statistical analysis Analysis of data was done by IBM computer using SPSS (statistical program for social science version 23): description of quantitative variables as Mean, SD, median and IQR, Shapiro test of normality used to check the data distribution, description of qualitative variables as number and percentage, Chi-square test was used to compare qualitative variables between groups, Fisher exact test was used when one expected cell or more are less than 5, Mann-Whitney test was used instead of unpaired t-test in non-parametric data (SD>30% mean). I considered the results statistically important when the important probability was less than 0.05 (P < 0.05). P-value < 0.001 was considered highly statistically important (HS), and P-value ≥ 0.05 was considered statistically insignificant (NS) (10).

ELIGIBILITY:
Inclusion Criteria:

* Patients with recurrent low output colo-cutaneous fistula (less than 500cc/24h) or leak after anterior resection due to rectal cancer

  * patients who subjected to conservative measures but failed
  * patient with good general condition (ASA I&II),
* patients with size of fistula less than 15mm
* patients with good nutritional status

Exclusion Criteria:

* patients with bad general condition (ASAIII&IV&V),
* patients with high output fistula ,
* patients with recto-vaginal or recto-vesical fistula,
* patients with size of fistula more than 15mm
* patients were treated with conservative measures.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2020-12-10 (Actual); Primary Completion 2022-05-10 (Actual); Study Completion 2022-08-10 (Actual)

PRIMARY OUTCOMES:
incidence of recurrence of fistula | within one week after the endoscopy
  incidence of recurrence of fistula

SECONDARY OUTCOMES:
incidence of side effects of endoscopy | within one month after the endoscopy
  incidence of side effects of endoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Said Mohamed Negm, Principal Investigator — Zagazig University Hospitals
Locations (1):
- Zagazig University Hospitals, Zagazig, Sharquia, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Negm S, Farag A, Shafiq A, Allah EA, Shehata M, Orban YA, Saleh M, Abdelghani AA. Endoscopic management of low output recurrent colonic fistula or leak after anterior resection for rectal cancer: a randomized controlled trial. Surg Endosc. 2023 Aug;37(8):6145-6152. doi: 10.1007/s00464-023-10092-z. Epub 2023 May 5. PMID 37145174